CLINICAL TRIAL: NCT04287218
Title: A Randomized Controlled Trial Comparing the Efficacy of Therapist Guided Internet-delivered Cognitive Therapy (TG-iConquerFear) With Augmented Treatment as Usual in Reducing Fear of Cancer Recurrence in Danish Colorectal Cancer Survivors
Brief Title: Reducing Fear of Cancer Recurrence in Danish Colorectal Cancer Survivors
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vejle Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Centre for Oncology Education and Research Translation (CONCERT), Australia (Unknown); Danish Cancer Society (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TG-iConquerFear
Record Dates: First submitted 2020-02-25; First posted 2020-02-27 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Fear of Cancer Recurrence; Colorectal Cancer; Anxiety; Health Anxiety; Bodily Distress Syndrome
Keywords: internet-based; digital health; cognitive therapy; randomized controlled trial
MeSH Terms: conditions — Colorectal Neoplasms; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Survey: The study is population based and cross sectional. Participants will be invited to complete an electronic questionnaire to screen for fear of cancer recurrence and other psychological factors.
  RCT: This part of the study is a population based, randomized, controlled clinical superiority trial. Participants are randomized to internet-based, therapist guided iConquerFear or augmented treatment as usual (1:1).
  If the planned number of participants (estimated by power calculation) has not been enrolled through the scheduled screening process, colorectal cancer survivors diagnosed during 2019 will be invited to the screening, and if needed, also colorectal cancer survivors diagnosed in 2020.
  The additional screening invitations will be sent out immediately after the last round of screening, i.e. before any follow-up data have been obtained. Hence, the statistical analyses will not be affected in any way.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TG-iConquerFear (Experimental): The participant is guided through the web-based sessions by minimum weekly contact with an experienced therapist (estimated ½ hour/week for 10 weeks). The therapist will motivate, answer questions and give feedback on written material and exercises.
  Interventions: Behavioral: TG-iConquerFear
- Augmented treatment as usual (Active Comparator): The control group is described as "augmented" treatment as usual (aTAU), since the diagnostic telephone interview exceeds standard treatment. Further more, the participants will be referred to a website with a non-guided, publicly available E-learning program in cancer rehabilitation hosted by the Region of Central Jutland (livogkraeft.rm.dk). In addition to written material the website includes self-help instructions for meditation.
  Interventions: Behavioral: aTAU

INTERVENTIONS:
Behavioral: TG-iConquerFear — The theoretical frame of iConquerFear is based on the Common-Sense Model of illness, the Self-Regulatory Executive Function model and Relational Frame Theory. The intervention includes elements of attention training, increasing metacognitive awareness, acceptance & mindfulness, promotion of appropriate screening behavior, and values-based goal setting. The electronic platform comprises 5 modules containing educational text, interactive exercises, short videos featuring doctors, therapists and patients' perspectives.
  Arms: TG-iConquerFear
Behavioral: aTAU — Active control group
  Other Names: Augmented treatment as usual
  Arms: Augmented treatment as usual

SUMMARY:
Cognitive therapy has been shown to reduce fear of cancer recurrence (FCR), mainly in breast cancer survivors. The accessibility of cognitive behavioural interventions could be further improved by Internet delivery, but self-guided interventions have shown limited efficacy. The aim of this study is to test the efficacy of a therapist guided internet-delivered intervention (TG-iConquerFear) vs. augmented treatment as usual (aTAU) in Danish colorectal cancer survivors.

DETAILED DESCRIPTION:
Colorectal cancer (CRC) screening, early detection, and improved treatment have led to rising survival rates over the past decades. This improvement has resulted in an increasing number of long-term CRC survivors with no residual disease. Most survivors manage to establish a 'new normal' after finishing treatment, but some survivors experience difficulties in normal functioning and decreased quality of life (QoL) due to substantial psychological strain. Anxiety and depression e.g. are reported in 34% of CRC survivors 1-5 years post-diagnosis. One of the most common concerns among cancer survivors is fear of cancer recurrence (FCR), defined as "Fear, worry or concern relating to the possibility that cancer will come back or progress". The severity of self-reported FCR does not seem to differ much according to cancer type and FCR can persist even among very long term survivors. Higher FCR is associated with multiple psychological factors including (health) anxiety, depression, greater uncertainty in illness, perceived risk of recurrence and negative beliefs about worry. An expert consensus on the defining features of clinical FCR suggested, that the following four features are key characteristics of clinical FCR: a) high levels of preoccupation; b) high levels of worry; c) that are persistent; and d) hypervigilance to bodily symptom.

Most CRC survivors report some degree of FCR. The term "clinically significant FCR" is introduced to describe when the strain of FCR becomes clinically important, negatively influencing the life of the survivor. Validated screening questionnaires, such as the Fear of Cancer Recurrence Inventory-Short Form (FCRI-SF), have been used to identify likely cases of clinically significant FCR. Two recent studies report likely clinically significant FCR based on the FCRI-SF among 13,7% and 10,1% of CRC survivors (unpublished data, personal communication with first authors). However, the prevalence of clinical FCR in CRC survivors is still somewhat uncertain, as estimates are based on small studies [n=51-91], or studies with simplistic or unvalidated FCR measures.

Two large cohort studies have focused on patient reported health-related QoL after (colorectal) cancer. The English study includes people "living with and beyond cancer", which does not distinguish between survivors with no residual disease, those living with cancer or with a history of recurrence. Furthermore, FCR is assessed with a single item. A Dutch study based on the PROFILES registry used the Impact of Cancer scale (Health Worries subscale) measure, which does not include a proposed cut-off score for clinical FCR. The current study will provide a more definitive estimate of the prevalence of clinical FCR in CRC survivors.

This study will also explore psychological factors related to FCR in CRC survivors. A cancer diagnosis is life changing and imposes heavy stress on patient and relatives. Together with often numerous physical symptoms and social changes after the cancer treatment, the net sum of stressors may exceed the cancer survivor's ability to adapt. This overload may manifest in the experience of bodily symptoms and in some cases develop into a functional disorder/somatic symptom disorder such as bodily distress syndrome or health anxiety, as proposed by Simonelli et al. Bodily distress syndrome is defined as a condition in which the patient suffers from, usually multiple, bodily symptoms in a characteristic pattern not attributable to verifiable, conventionally defined diseases.

Health anxiety is characterized by preoccupation with fear of having a serious and life-threatening illness with no objective sign of disease, which persists despite medical reassurance. Health anxiety and FCR overlap somewhat, as they both include unpleasant thoughts or ruminations, which interfere with everyday life and may lead to further unnecessary investigations and treatments. One study investigated hypochondriasis in breast cancer survivors and found that 43% of those with a clinical level of FCR met the diagnostic criteria. Two studies of one CRC cohort have measured somatization (i.e. manifestation of physiological distress as physical symptoms), but not links with FCR. To the best of our knowledge, no previous studies have investigated the relationship between functional disorders, FCR, anxiety and depression in CRC survivors.

Illness uncertainty has been linked with FCR and health anxiety. When diagnosed asymptomatic through screening, illness uncertainty might by heightened. Therefore, diagnosis via screening may lead to increased issues in coping with the cancer and FCR. The comprehensive Danish Clinical Cancer Registries contain data on the method of diagnosis, namely whether the CRC survivor was diagnosed through the Danish nationwide Colorectal Cancer Screening Program, as opposed to diagnosed as a result of symptoms. This enables research in this unexplored area of psychosocial consequences of screen-detected cancers.

Around one fourth (26,5%) of CRC survivors and 20-56% of people living with and beyond CRC report psychosocial assistance in coping with FCR to be an important unmet need. Randomized controlled trials testing interventions for reducing FCR have primarily been conducted in breast or mixed cancer survivor populations. Most interventions are based on variations of cognitive-behavioural therapy (CBT). Contemporary CBTs aiming to modify cognitive processes (e.g., attentional bias and beliefs about worry) rather than thought content (e.g. thoughts of death) were more effective (g=0.42 vs 0.24). The delivery format of interventions previously or currently being evaluated has been group, face-to-face, blended, by telephone or by web-based platforms.

"ConquerFear" is an individual face-to-face therapist-delivered intervention with demonstrated efficacy in reducing FCR compared to a relaxation training attention control group of patients with mixed cancers of whom the majority (89%) were women with breast cancer. While use of ConquerFear has been sustained by many study therapists beyond the end of the study, it is a resource and time-consuming approach accessible primarily to those in close proximity to major metropolitan cancer centres with highly trained psychologists. Consequently, a web-based self-management version of ConquerFear has been created (iConquerFear), similar in curriculum content but different in delivery. Qualitative evaluation of the usability of iConquerFear showed: iConquerFear was normalising and empowering; flexible access was key; delivery mode was engaging; tailoring was crucial; links to additional resources were valued.

Web-based interventions have the potential to fill an important gap in quality cancer care by augmenting limited available mental health services. However, there is some evidence that entirely self-guided web-based FCR interventions may have limited efficacy, and it has been suggested that therapist input may increase efficacy. Web-based therapist-guided cognitive therapy has advantages for both patients and providers and effects appear comparable to traditional face-to-face therapy in treating distress in patients with cancer. Evidence suggests that guided web-based interventions are superior to unguided interventions.

Aim The primary aim of this RCT is to test if a therapist-guided version of iConquerFear (TG-iConquerFear) can reduce FCR and improve QoL for CRC survivors more than augmented treatment as usual (aTAU).

Secondary objectives are to i) outline the prevalence of FCR in a population based CRC cohort up to 5 years post-diagnosis using a validated FCR measure with a clinical cut-off. This comprehensive screening will also be used to recruit to the RCT of TG-iConquerFear.

ii) outline the prevalence of anxiety, depression, bodily distress syndrome and health anxiety in a population based CRC cohort up to 5 years post-diagnosis.

iii) investigate whether being diagnosed as a consequence of the Danish Nation-wide Colorectal Cancer Screening Program increases FCR compared to being diagnosed based on physical symptoms and whether this relationship is mediated by increased uncertainty in illness.

iv) investigate whether FCR is associated with anxiety, depression, bodily distress syndrome and health anxiety in CRC survivors, as well as investigate whether uncertainty in illness, negative beliefs about worry and perceived risk of cancer recurrence act as moderators or mediators of these relationships.

v) examine the cost-effectiveness of the TG-iConquerFear intervention versus aTAU.

ELIGIBILITY:
Inclusion Criteria:

* Completed curative intent colorectal cancer treatment with surgery and/or radiation and/or adjuvant chemotherapy between 1 March 2014 and 31 December 2018
* No history of recurrence after primary operation
* Fear of Cancer Recurrence Inventory score of 22 or above (14)
* Age 18 or above
* Reads and understands Danish
* Access and ability to use Internet

Exclusion Criteria:

* Cancer recurrence at any follow-up
* Inability to comply with the protocol due to severe psychiatric, cognitive disorder or substance abuse identified during telephone interview
* As the intervention is web-based, participants without knowledge of or access to the Internet will be excluded from the RCT (including dyslexia).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-05-10 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change of total score on Fear of Cancer Recurrence Inventory (FCRI) from baseline to 2nd follow-up | 3 months post-intervention
  Questionnaire

SECONDARY OUTCOMES:
Change of total score on Fear of Cancer Recurrence Inventory (FCRI) from baseline | 1-14 days after intervention and after 6 and 12 months
  Questionnaire
Change in Bodily Distress Syndrome from baseline as evaluated by the BDS Checklist | 1-14 days after intervention and after 6 and 12 months
  Questionnaire
Change in anxiety and depression from baseline as evaluated by the relevant Symptom Checklist-90-R | 1-14 days after intervention and after 6 and 12 months
  Questionnaire
Change in health anxiety from baseline as measured by the Whiteley-6 index | 1-14 days after intervention and after 6 and 12 months
  Questionnaire
Evaluation of cost-effectiveness of TG-iConquerFear | Max. 27 months
  Information will be extracted from Danish registries.
Comparison of changes in health care usage between intervention arm and aTAU | Max. 27 months
  Information will be extracted from Danish registries.

OTHER OUTCOMES:
Change in uncertainty in illness as evaluated by Mishels Uncertainty of Illness Scale (MUIS). | Twice during the intervention, 1-14 days after the intervention and after 3, 6, and 12 months
  Process measures. Questionnaire
Change of negative beliefs about worry evaluated by MetaCognitions Questionnaire-30. | Twice during the intervention, 1-14 days after the intervention and after 3, 6, and 12 months
  Process measures. Questionnaire
Perceived risk of recurrence measured by the visual analogue scale from 1-100 | Twice during the intervention, 1-14 days after the intervention and after 3, 6, and 12 months
  Process measures. Scale.

CONTACTS AND LOCATIONS:
Overall Officials: Lars Henrik Jensen, MD, PhD, Study Chair — Vejle Hospital
Locations (1):
- Vejle Hospital, University Hospital of Southern Denmark, Vejle, Denmark

IPD SHARING:
Plan to Share IPD: No
Data will be available up on request

REFERENCES:
- [Background] Jefford M, Ward AC, Lisy K, Lacey K, Emery JD, Glaser AW, Cross H, Krishnasamy M, McLachlan SA, Bishop J. Patient-reported outcomes in cancer survivors: a population-wide cross-sectional study. Support Care Cancer. 2017 Oct;25(10):3171-3179. doi: 10.1007/s00520-017-3725-5. Epub 2017 Apr 22. PMID 28434095
- [Background] Simard S, Thewes B, Humphris G, Dixon M, Hayden C, Mireskandari S, Ozakinci G. Fear of cancer recurrence in adult cancer survivors: a systematic review of quantitative studies. J Cancer Surviv. 2013 Sep;7(3):300-22. doi: 10.1007/s11764-013-0272-z. Epub 2013 Mar 10. PMID 23475398
- [Background] Lebel S, Ozakinci G, Humphris G, Mutsaers B, Thewes B, Prins J, Dinkel A, Butow P; University of Ottawa Fear of Cancer Recurrence Colloquium attendees. From normal response to clinical problem: definition and clinical features of fear of cancer recurrence. Support Care Cancer. 2016 Aug;24(8):3265-8. doi: 10.1007/s00520-016-3272-5. Epub 2016 May 12. PMID 27169703
- [Background] van de Wal M, van de Poll-Franse L, Prins J, Gielissen M. Does fear of cancer recurrence differ between cancer types? A study from the population-based PROFILES registry. Psychooncology. 2016 Jul;25(7):772-8. doi: 10.1002/pon.4002. Epub 2015 Oct 14. PMID 26464337
- [Background] Koch L, Jansen L, Brenner H, Arndt V. Fear of recurrence and disease progression in long-term (>/= 5 years) cancer survivors--a systematic review of quantitative studies. Psychooncology. 2013 Jan;22(1):1-11. doi: 10.1002/pon.3022. Epub 2012 Jan 10. PMID 22232030
- [Background] McGinty HL, Small BJ, Laronga C, Jacobsen PB. Predictors and patterns of fear of cancer recurrence in breast cancer survivors. Health Psychol. 2016 Jan;35(1):1-9. doi: 10.1037/hea0000238. Epub 2015 Jun 1. PMID 26030308
- [Background] Deimling GT, Bowman KF, Sterns S, Wagner LJ, Kahana B. Cancer-related health worries and psychological distress among older adult, long-term cancer survivors. Psychooncology. 2006 Apr;15(4):306-20. doi: 10.1002/pon.955. PMID 16041841
- [Background] Smith A', Sharpe L, Thewes B, Turner J, Gilchrist J, Fardell JE, Girgis A, Tesson S, Descallar J, Bell ML, Beith J, Butow P; ConquerFear Authorship Group. Medical, demographic and psychological correlates of fear of cancer recurrence (FCR) morbidity in breast, colorectal and melanoma cancer survivors with probable clinically significant FCR seeking psychological treatment through the ConquerFear study. Support Care Cancer. 2018 Dec;26(12):4207-4216. doi: 10.1007/s00520-018-4294-y. Epub 2018 Jun 7. PMID 29882025
- [Background] Mutsaers B, Butow P, Dinkel A, Humphris G, Maheu C, Ozakinci G, Prins J, Sharpe L, Smith AB, Thewes B, Lebel S. Identifying the key characteristics of clinical fear of cancer recurrence: An international Delphi study. Psychooncology. 2020 Feb;29(2):430-436. doi: 10.1002/pon.5283. Epub 2019 Nov 25. PMID 31713279
- [Background] Waters EA, Arora NK, Klein WM, Han PK. Perceived risk, trust and health-related quality of life among cancer survivors. Ann Behav Med. 2010 Feb;39(1):91-7. doi: 10.1007/s12160-010-9163-y. PMID 20333563
- [Background] Mullens AB, McCaul KD, Erickson SC, Sandgren AK. Coping after cancer: risk perceptions, worry, and health behaviors among colorectal cancer survivors. Psychooncology. 2004 Jun;13(6):367-76. doi: 10.1002/pon.751. PMID 15188444
- [Background] Steele N, Haigh R, Knowles G, Mackean M. Carcinoembryonic antigen (CEA) testing in colorectal cancer follow up: what do patients think? Postgrad Med J. 2007 Sep;83(983):612-4. doi: 10.1136/pgmj.2007.059634. PMID 17823231
- [Background] Fisher A, Beeken RJ, Heinrich M, Williams K, Wardle J. Health behaviours and fear of cancer recurrence in 10 969 colorectal cancer (CRC) patients. Psychooncology. 2016 Dec;25(12):1434-1440. doi: 10.1002/pon.4076. Epub 2016 Feb 11. PMID 26863926
- [Background] Fardell JE, Jones G, Smith AB, Lebel S, Thewes B, Costa D, Tiller K, Simard S, Feldstain A, Beattie S, McCallum M; Conquer Fear authorship group; Butow P. Exploring the screening capacity of the Fear of Cancer Recurrence Inventory-Short Form for clinical levels of fear of cancer recurrence. Psychooncology. 2018 Feb;27(2):492-499. doi: 10.1002/pon.4516. Epub 2017 Aug 18. PMID 28755462
- [Background] Simard S, Savard J. Fear of Cancer Recurrence Inventory: development and initial validation of a multidimensional measure of fear of cancer recurrence. Support Care Cancer. 2009 Mar;17(3):241-51. doi: 10.1007/s00520-008-0444-y. Epub 2008 Apr 15. PMID 18414902
- [Background] Hovdenak Jakobsen I, Jeppesen MM, Simard S, Thaysen HV, Laurberg S, Juul T. Initial validation of the Danish version of the Fear of Cancer Recurrence Inventory (FCRI) in colorectal cancer patients. J Cancer Surviv. 2018 Dec;12(6):723-732. doi: 10.1007/s11764-018-0709-5. Epub 2018 Aug 20. PMID 30128857
- [Background] Custers JAE, Gielissen MFM, Janssen SHV, de Wilt JHW, Prins JB. Fear of cancer recurrence in colorectal cancer survivors. Support Care Cancer. 2016 Feb;24(2):555-562. doi: 10.1007/s00520-015-2808-4. Epub 2015 Jun 25. PMID 26108170
- [Background] Glaser AW, Fraser LK, Corner J, Feltbower R, Morris EJ, Hartwell G, Richards M, Wagland R. Patient-reported outcomes of cancer survivors in England 1-5 years after diagnosis: a cross-sectional survey. BMJ Open. 2013 Apr 10;3(4):e002317. doi: 10.1136/bmjopen-2012-002317. Print 2013. PMID 23578682
- [Background] Downing A, Morris EJ, Richards M, Corner J, Wright P, Sebag-Montefiore D, Finan P, Kind P, Wood C, Lawton S, Feltbower R, Wagland R, Vernon S, Thomas J, Glaser AW. Health-related quality of life after colorectal cancer in England: a patient-reported outcomes study of individuals 12 to 36 months after diagnosis. J Clin Oncol. 2015 Feb 20;33(6):616-24. doi: 10.1200/JCO.2014.56.6539. Epub 2015 Jan 5. PMID 25559806
- [Background] Simonelli LE, Siegel SD, Duffy NM. Fear of cancer recurrence: a theoretical review and its relevance for clinical presentation and management. Psychooncology. 2017 Oct;26(10):1444-1454. doi: 10.1002/pon.4168. Epub 2016 Jun 1. PMID 27246348
- [Background] Fink P, Schroder A. One single diagnosis, bodily distress syndrome, succeeded to capture 10 diagnostic categories of functional somatic syndromes and somatoform disorders. J Psychosom Res. 2010 May;68(5):415-26. doi: 10.1016/j.jpsychores.2010.02.004. PMID 20403500
- [Background] Tyrer P, Eilenberg T, Fink P, Hedman E, Tyrer H. Health anxiety: the silent, disabling epidemic. BMJ. 2016 Apr 25;353:i2250. doi: 10.1136/bmj.i2250. No abstract available. PMID 27112356
- [Background] Fink P, Ornbol E, Toft T, Sparle KC, Frostholm L, Olesen F. A new, empirically established hypochondriasis diagnosis. Am J Psychiatry. 2004 Sep;161(9):1680-91. doi: 10.1176/appi.ajp.161.9.1680. PMID 15337660
- [Background] Thewes B, Bell ML, Butow P, Beith J, Boyle F, Friedlander M, McLachlan SA; Members of the FCR Study Advisory Committee. Psychological morbidity and stress but not social factors influence level of fear of cancer recurrence in young women with early breast cancer: results of a cross-sectional study. Psychooncology. 2013 Dec;22(12):2797-806. doi: 10.1002/pon.3348. Epub 2013 Aug 23. PMID 24038525
- [Background] Chambers SK, Baade P, Meng X, Youl P, Aitken J, Dunn J. Survivor identity after colorectal cancer: antecedents, prevalence and outcomes. Psychooncology. 2012 Sep;21(9):962-9. doi: 10.1002/pon.1991. Epub 2011 May 24. PMID 21608073
- [Background] Dunn J, Ng SK, Holland J, Aitken J, Youl P, Baade PD, Chambers SK. Trajectories of psychological distress after colorectal cancer. Psychooncology. 2013 Aug;22(8):1759-65. doi: 10.1002/pon.3210. Epub 2012 Nov 5. PMID 23125004
- [Background] Lebel S, Maheu C, Tomei C, Bernstein LJ, Courbasson C, Ferguson S, Harris C, Jolicoeur L, Lefebvre M, Muraca L, Ramanakumar AV, Singh M, Parrott J, Figueiredo D. Towards the validation of a new, blended theoretical model of fear of cancer recurrence. Psychooncology. 2018 Nov;27(11):2594-2601. doi: 10.1002/pon.4880. Epub 2018 Sep 27. PMID 30180279
- [Background] Eilenberg T, Kronstrand L, Fink P, Frostholm L. Acceptance and commitment group therapy for health anxiety--results from a pilot study. J Anxiety Disord. 2013 Jun;27(5):461-8. doi: 10.1016/j.janxdis.2013.06.001. Epub 2013 Jun 19. PMID 23871841
- [Background] Kotronoulas G, Papadopoulou C, Burns-Cunningham K, Simpson M, Maguire R. A systematic review of the supportive care needs of people living with and beyond cancer of the colon and/or rectum. Eur J Oncol Nurs. 2017 Aug;29:60-70. doi: 10.1016/j.ejon.2017.05.004. Epub 2017 May 30. PMID 28720267
- [Background] Tauber NM, O'Toole MS, Dinkel A, Galica J, Humphris G, Lebel S, Maheu C, Ozakinci G, Prins J, Sharpe L, Smith AB, Thewes B, Simard S, Zachariae R. Effect of Psychological Intervention on Fear of Cancer Recurrence: A Systematic Review and Meta-Analysis. J Clin Oncol. 2019 Nov 1;37(31):2899-2915. doi: 10.1200/JCO.19.00572. Epub 2019 Sep 18. PMID 31532725
- [Background] Herschbach P, Book K, Dinkel A, Berg P, Waadt S, Duran G, Engst-Hastreiter U, Henrich G. Evaluation of two group therapies to reduce fear of progression in cancer patients. Support Care Cancer. 2010 Apr;18(4):471-9. doi: 10.1007/s00520-009-0696-1. Epub 2009 Oct 29. PMID 19865833
- [Background] Maheu C, Lebel S, Courbasson C, Lefebvre M, Singh M, Bernstein LJ, Muraca L, Benea A, Jolicoeur L, Harris C, Ramanakumar AV, Ferguson S, Sidani S. Protocol of a randomized controlled trial of the fear of recurrence therapy (FORT) intervention for women with breast or gynecological cancer. BMC Cancer. 2016 Apr 25;16:291. doi: 10.1186/s12885-016-2326-x. PMID 27112319
- [Background] Merckaert I, Lewis F, Delevallez F, Herman S, Caillier M, Delvaux N, Libert Y, Lienard A, Nogaret JM, Ogez D, Scalliet P, Slachmuylder JL, Van Houtte P, Razavi D. Improving anxiety regulation in patients with breast cancer at the beginning of the survivorship period: a randomized clinical trial comparing the benefits of single-component and multiple-component group interventions. Psychooncology. 2017 Aug;26(8):1147-1154. doi: 10.1002/pon.4294. Epub 2016 Nov 7. PMID 27718533
- [Background] Butow PN, Turner J, Gilchrist J, Sharpe L, Smith AB, Fardell JE, Tesson S, O'Connell R, Girgis A, Gebski VJ, Asher R, Mihalopoulos C, Bell ML, Zola KG, Beith J, Thewes B. Randomized Trial of ConquerFear: A Novel, Theoretically Based Psychosocial Intervention for Fear of Cancer Recurrence. J Clin Oncol. 2017 Dec 20;35(36):4066-4077. doi: 10.1200/JCO.2017.73.1257. Epub 2017 Nov 2. PMID 29095681
- [Background] Tomei C, Lebel S, Maheu C, Lefebvre M, Harris C. Examining the preliminary efficacy of an intervention for fear of cancer recurrence in female cancer survivors: a randomized controlled clinical trial pilot study. Support Care Cancer. 2018 Aug;26(8):2751-2762. doi: 10.1007/s00520-018-4097-1. Epub 2018 Mar 2. PMID 29500582
- [Background] Davidson J, Malloch M, Humphris G. A single-session intervention (the Mini-AFTERc) for fear of cancer recurrence: A feasibility study. Psychooncology. 2018 Nov;27(11):2668-2670. doi: 10.1002/pon.4724. Epub 2018 Apr 30. No abstract available. PMID 29624779
- [Background] van de Wal M, Thewes B, Gielissen M, Speckens A, Prins J. Efficacy of Blended Cognitive Behavior Therapy for High Fear of Recurrence in Breast, Prostate, and Colorectal Cancer Survivors: The SWORD Study, a Randomized Controlled Trial. J Clin Oncol. 2017 Jul 1;35(19):2173-2183. doi: 10.1200/JCO.2016.70.5301. Epub 2017 May 4. PMID 28471726
- [Background] Cruickshank S, Steel E, Fenlon D, Armes J, Scanlon K, Banks E, Humphris G. A feasibility study of the Mini-AFTER telephone intervention for the management of fear of recurrence in breast cancer survivors: a mixed-methods study protocol. Pilot Feasibility Stud. 2017 Jul 20;4:22. doi: 10.1186/s40814-017-0161-8. eCollection 2018. PMID 28748105
- [Background] Dieng M, Butow PN, Costa DS, Morton RL, Menzies SW, Mireskandari S, Tesson S, Mann GJ, Cust AE, Kasparian NA. Psychoeducational Intervention to Reduce Fear of Cancer Recurrence in People at High Risk of Developing Another Primary Melanoma: Results of a Randomized Controlled Trial. J Clin Oncol. 2016 Dec 20;34(36):4405-4414. doi: 10.1200/JCO.2016.68.2278. Epub 2016 Oct 28. PMID 27998215
- [Background] van Helmondt SJ, van der Lee ML, de Vries J. Study protocol of the CAREST-trial: a randomised controlled trial on the (cost-) effectiveness of a CBT-based online self-help training for fear of cancer recurrence in women with curatively treated breast cancer. BMC Cancer. 2016 Jul 25;16:527. doi: 10.1186/s12885-016-2562-0. PMID 27455846
- [Background] Murphy MJ, Newby JM, Butow P, Kirsten L, Allison K, Loughnan S, Price MA, Shaw J, Shepherd H, Smith J, Andrews G. iCanADAPT Early protocol: randomised controlled trial (RCT) of clinician supervised transdiagnostic internet-delivered cognitive behaviour therapy (iCBT) for depression and/or anxiety in early stage cancer survivors -vs- treatment as usual. BMC Cancer. 2017 Mar 15;17(1):193. doi: 10.1186/s12885-017-3182-z. PMID 28298187
- [Background] Willems RA, Bolman CA, Mesters I, Kanera IM, Beaulen AA, Lechner L. Cancer survivors in the first year after treatment: the prevalence and correlates of unmet needs in different domains. Psychooncology. 2016 Jan;25(1):51-7. doi: 10.1002/pon.3870. Epub 2015 Jun 25. PMID 26110652
- [Background] Butow P, Williams D, Thewes B, Tesson S, Sharpe L, Smith AB, Fardell JE, Turner J, Gilchrist J, Girgis A, Beith J; Conquer Fear Authorship Group. A psychological intervention (ConquerFear) for treating fear of cancer recurrence: Views of study therapists regarding sustainability. Psychooncology. 2019 Mar;28(3):533-539. doi: 10.1002/pon.4971. Epub 2019 Jan 15. PMID 30597658
- [Background] Smith AB, Bamgboje-Ayodele A, Butow P, Klein B, Turner J, Sharpe L, Fardell J, Beatty L, Pearce A, Thewes B, Beith J; iConquerFear Community Advisory Group; Girgis A. Development and usability evaluation of an online self-management intervention for fear of cancer recurrence (iConquerFear). Psychooncology. 2020 Jan;29(1):98-106. doi: 10.1002/pon.5218. Epub 2019 Sep 10. PMID 31483911
- [Background] Leykin Y, Thekdi SM, Shumay DM, Munoz RF, Riba M, Dunn LB. Internet interventions for improving psychological well-being in psycho-oncology: review and recommendations. Psychooncology. 2012 Sep;21(9):1016-25. doi: 10.1002/pon.1993. Epub 2011 May 24. PMID 21608075
- [Background] van Helmondt SJ, van der Lee ML, van Woezik RAM, Lodder P, de Vries J. No effect of CBT-based online self-help training to reduce fear of cancer recurrence: First results of the CAREST multicenter randomized controlled trial. Psychooncology. 2020 Jan;29(1):86-97. doi: 10.1002/pon.5233. Epub 2019 Nov 13. PMID 31595627
- [Background] Compen F, Bisseling E, Schellekens M, Donders R, Carlson L, van der Lee M, Speckens A. Face-to-Face and Internet-Based Mindfulness-Based Cognitive Therapy Compared With Treatment as Usual in Reducing Psychological Distress in Patients With Cancer: A Multicenter Randomized Controlled Trial. J Clin Oncol. 2018 Aug 10;36(23):2413-2421. doi: 10.1200/JCO.2017.76.5669. Epub 2018 Jun 28. PMID 29953304
- [Background] Spek V, Cuijpers P, Nyklicek I, Riper H, Keyzer J, Pop V. Internet-based cognitive behaviour therapy for symptoms of depression and anxiety: a meta-analysis. Psychol Med. 2007 Mar;37(3):319-28. doi: 10.1017/S0033291706008944. Epub 2006 Nov 20. PMID 17112400
- [Background] Pihlaja S, Stenberg JH, Joutsenniemi K, Mehik H, Ritola V, Joffe G. Therapeutic alliance in guided internet therapy programs for depression and anxiety disorders - A systematic review. Internet Interv. 2017 Nov 17;11:1-10. doi: 10.1016/j.invent.2017.11.005. eCollection 2018 Mar. PMID 30135754
- [Background] Beaton DE, Bombardier C, Guillemin F, Ferraz MB. Guidelines for the process of cross-cultural adaptation of self-report measures. Spine (Phila Pa 1976). 2000 Dec 15;25(24):3186-91. doi: 10.1097/00007632-200012150-00014. No abstract available. PMID 11124735
- [Background] McMullen C, Bulkley J, Corley DA, Madrid S, Davis AQ, Hesselbrock R, Kurtilla F, Anderson CK, Arterburn D, Somkin CP, Pawloski PA, Ghai NR, Feigelson HS. Health care improvement and survivorship priorities of colorectal cancer survivors: findings from the PORTAL colorectal cancer cohort survey. Support Care Cancer. 2019 Jan;27(1):147-156. doi: 10.1007/s00520-018-4299-6. Epub 2018 Jun 12. PMID 29948396
- [Background] Chan AW, Tetzlaff JM, Gotzsche PC, Altman DG, Mann H, Berlin JA, Dickersin K, Hrobjartsson A, Schulz KF, Parulekar WR, Krleza-Jeric K, Laupacis A, Moher D. SPIRIT 2013 explanation and elaboration: guidance for protocols of clinical trials. BMJ. 2013 Jan 8;346:e7586. doi: 10.1136/bmj.e7586. PMID 23303884
- [Background] Nienhuis FJ, van de Willige G, Rijnders CA, de Jonge P, Wiersma D. Validity of a short clinical interview for psychiatric diagnosis: the mini-SCAN. Br J Psychiatry. 2010 Jan;196(1):64-8. doi: 10.1192/bjp.bp.109.066563. PMID 20044664
- [Background] Petersen MW, Schroder A, Jorgensen T, Ornbol E, Dantoft TM, Eliasen M, Fink P. RIFD - A brief clinical research interview for functional somatic disorders and health anxiety. J Psychosom Res. 2019 Jul;122:104-111. doi: 10.1016/j.jpsychores.2019.04.001. Epub 2019 Apr 2. PMID 30955913
- [Background] Short CE, DeSmet A, Woods C, Williams SL, Maher C, Middelweerd A, Muller AM, Wark PA, Vandelanotte C, Poppe L, Hingle MD, Crutzen R. Measuring Engagement in eHealth and mHealth Behavior Change Interventions: Viewpoint of Methodologies. J Med Internet Res. 2018 Nov 16;20(11):e292. doi: 10.2196/jmir.9397. PMID 30446482
- [Background] Lebel S, Simard S, Harris C, Feldstain A, Beattie S, McCallum M, Lefebvre M, Savard J, Devins GM. Empirical validation of the English version of the Fear of Cancer Recurrence Inventory. Qual Life Res. 2016 Feb;25(2):311-321. doi: 10.1007/s11136-015-1088-2. Epub 2015 Sep 4. PMID 26341969
- [Background] Costa DSJ, Smith AB, Fardell JE. The sum of all fears: conceptual challenges with measuring fear of cancer recurrence. Support Care Cancer. 2016 Jan;24(1):1-3. doi: 10.1007/s00520-015-2943-y. Epub 2015 Sep 16. PMID 26377307
- [Background] Costa DSJ. Screening for clinical levels of fear of cancer recurrence. Psychooncology. 2017 Nov;26(11):2002-2003. doi: 10.1002/pon.4390. Epub 2017 Feb 10. No abstract available. PMID 28146299
- [Background] Budtz-Lilly A, Fink P, Ornbol E, Vestergaard M, Moth G, Christensen KS, Rosendal M. A new questionnaire to identify bodily distress in primary care: The 'BDS checklist'. J Psychosom Res. 2015 Jun;78(6):536-45. doi: 10.1016/j.jpsychores.2015.03.006. Epub 2015 Mar 16. PMID 25818346
- [Background] PARLOFF MB, KELMAN HC, FRANK JD. Comfort, effectiveness, and self-awareness as criteria of improvement in psychotherapy. Am J Psychiatry. 1954 Nov;111(5):343-52. doi: 10.1176/ajp.111.5.343. No abstract available. PMID 13197596
- [Background] Fink P, Ewald H, Jensen J, Sorensen L, Engberg M, Holm M, Munk-Jorgensen P. Screening for somatization and hypochondriasis in primary care and neurological in-patients: a seven-item scale for hypochondriasis and somatization. J Psychosom Res. 1999 Mar;46(3):261-73. doi: 10.1016/s0022-3999(98)00092-0. PMID 10193917
- [Background] Veddegjaerde KE, Sivertsen B, Wilhelmsen I, Skogen JC. Confirmatory factor analysis and item response theory analysis of the Whiteley Index. Results from a large population based study in Norway. The Hordaland Health Study (HUSK). J Psychosom Res. 2014 Sep;77(3):213-8. doi: 10.1016/j.jpsychores.2014.06.011. Epub 2014 Jun 28. PMID 25149031
- [Background] Mishel MH. The measurement of uncertainty in illness. Nurs Res. 1981 Sep-Oct;30(5):258-63. PMID 6912987
- [Background] Hagen KB, Aas T, Lode K, Gjerde J, Lien E, Kvaloy JT, Lash TL, Soiland H, Lind R. Illness uncertainty in breast cancer patients: validation of the 5-item short form of the Mishel Uncertainty in Illness Scale. Eur J Oncol Nurs. 2015 Apr;19(2):113-9. doi: 10.1016/j.ejon.2014.10.009. Epub 2014 Dec 20. PMID 25538036
- [Background] Wells A, Cartwright-Hatton S. A short form of the metacognitions questionnaire: properties of the MCQ-30. Behav Res Ther. 2004 Apr;42(4):385-96. doi: 10.1016/S0005-7967(03)00147-5. PMID 14998733
- [Background] Cartwright-Hatton S, Wells A. Beliefs about worry and intrusions: the Meta-Cognitions Questionnaire and its correlates. J Anxiety Disord. 1997 May-Jun;11(3):279-96. doi: 10.1016/s0887-6185(97)00011-x. PMID 9220301
- [Derived] Lyhne JD, Smith AB, Timm S, Klein B, Thewes B, Girgis A, Bamgboje-Ayodele A, Beatty L, Fardell J, Fink P, Butow P, Frostholm L, Jensen LH. E-Health Intervention for Fear of Cancer Recurrence: A Randomized Clinical Trial. JAMA Netw Open. 2025 Nov 3;8(11):e2542112. doi: 10.1001/jamanetworkopen.2025.42112. PMID 41217757
- [Derived] Lyhne JD, Smith A'B, Frostholm L, Fink P, Jensen LH. Study protocol: a randomized controlled trial comparing the efficacy of therapist guided internet-delivered cognitive therapy (TG-iConquerFear) with augmented treatment as usual in reducing fear of cancer recurrence in Danish colorectal cancer survivors. BMC Cancer. 2020 Mar 16;20(1):223. doi: 10.1186/s12885-020-06731-6. PMID 32178640